CLINICAL TRIAL: NCT02537496
Title: Enhancing Working Memory in Patients With Early Alzheimer's Disease Through the Enhancement of Dorsolateral Prefrontal Cortex Neuroplasticity: A TMS-EEG Study
Brief Title: Enhancing Working Memory in Patients With Early Alzheimer's Disease Through the Use of rTMS
Acronym: rTMS-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Brain & Behavior Research Foundation (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Sanjeev Kumar, Sanjeev Kumar, MD, FRCPC, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 005/2015
Record Dates: First submitted 2015-07-30; First posted 2015-09-01 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Brain stimulation; Transcranial Magnetic Stimulation; Neuroplasticity; cognitive enhancement; TMS-EEG; rTMS; PAS
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be assigned randomly to a 4-week repetitive course of either rTMS or control intervention (Sham rTMS) that is similar to rTMS but does not produce the same amount of brain stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active placebo coil will be used as a Sham condition. This coil effectively mimics the real stimulation producing somatic sensation and sound (contraction of scalp muscles) with minimal direct brain effects. Same stimulation parameters and site as active condition will be used.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alzheimer's disease rTMS (Experimental): The intervention procedure done in this group is repetitive Transcranial Magnetic Stimulation.
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation
- Alzheimer's disease rTMS Sham (Sham Comparator): The intervention procedure done in this group is Repetitive Transcranial Magnetic Stimulation - Sham
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation - Sham
- Healthy Control (No Intervention): Healthy control group will only participate in baseline assessments which include baseline neuropsychological testing and baseline measurement of neuroplasticity. This will be used to standardize neuropsychological test scores and to compare the baseline neuroplasticity between healthy participants and Alzheimer's disease (AD) participants. Healthy control group will not get rTMS intervention.

INTERVENTIONS:
Procedure: Repetitive Transcranial Magnetic Stimulation — Active treatment will be delivered at 90% resting motor threshold intensity. Stimulation will be administered at 20 Hz with 25 stimulation trains of 30 stimuli each with an inter-train interval of 30 sec. Treatment will be applied in sequential order bilaterally to the left and right DLPFC.
  Other Names: rTMS
  Arms: Alzheimer's disease rTMS
Procedure: Repetitive Transcranial Magnetic Stimulation - Sham — Same stimulation parameters and site as active condition will be used, but with placebo coil which will have minimal direct brain effects
  Other Names: rTMS - Sham
  Arms: Alzheimer's disease rTMS Sham

SUMMARY:
In this study the investigators aim at assessing and then enhancing neuroplasticity in the dorsolateral prefrontal cortex (DLPFC) and working memory - a key function of DLPFC - in patients with mild Alzheimer's disease (AD). The investigators will use Paired Associative Stimulation (PAS) paradigm to measure neuroplasticity and then a 4-week course of high-frequency repetitive Transcranial Magnetic Stimulation (rTMS) to the DLPFC to enhance cognitive function. Clinical and cognitive assessments will be done at baseline, one week, one month and 6 months after the rTMS course. Healthy controls will also be enrolled to carry out baseline cognitive assessments and a baseline measurement of neuroplasticity.

DETAILED DESCRIPTION:
Specific aim 1: To assess working memory in participants with Alzheimer's disease (AD) and its change in response to a 4-week course of bilateral rTMS of DLPFC.

Hypothesis 1a: Compared to healthy individuals, participants with AD will be impaired on the N-back task.

Hypothesis 1b: Compared to sham rTMS, active rTMS will result in improvement on the N-back task in participants with AD at 1 week and 4 weeks after the treatment.

Specific aim 2: To assess DLPFC theta-gamma coupling during working memory performance in AD and its change in response to a 4-week course of bilateral rTMS of DLPFC.

Hypothesis 2a: Compared to healthy individuals, participants with AD will be impaired on DLPFC theta-gamma coupling during the N-back task.

Hypothesis 2b & 2c: Compared to sham rTMS, active rTMS will result in improvement in DLPFC theta-gamma coupling during the N-back task in participants with AD at 1 week and 4 weeks after the treatment.

Specific aim 3: To assess DLPFC neuroplasticity using PAS in participants with AD and its change in response to a 4-week course of bilateral rTMS.

Hypothesis 3a: Compared to healthy individuals, participants with AD will be impaired on PAS-induced neuroplasticity.

Hypothesis 3b: Compared to sham rTMS, active rTMS will result in improvement on PAS-induced neuroplasticity in participants with AD at 1 week and 4 weeks after the treatment.

Specific aim 4: To assess change in working memory, theta gamma coupling and DLPFC neuroplasticity at 6 months after the course of bilateral rTMS.

Hypothesis 4: Compared to sham rTMS, active rTMS group will perform better on measures of working memory, theta gamma coupling and PAS- induced DLPFC neuroplasticity 6 months after the course of rTMS.

Specific aim 5: To assess the change in general cognitive function at 4 weeks and 6 months after the course of bilateral rTMS.

Hypothesis 5: Compared to sham rTMS, active rTMS group will perform better on measures of general cognitive function at 4 weeks and 6 months after the course of rTMS.

Specific Aim 6: To assess insight in AD at baseline and any change in insight at 4 week and 6 month post rTMS follow up. H6: Participants with AD will have impaired insight into illness and cognitive function and they will experience improved insight at 4 week and 6 month follow up points.

Specific Aim 7: To validate a new scale for insight in AD , 'The Scale to Assess Anosognosia in Neurocognitive Disorders' (SAND) for its ability to assess insight at baseline and any change at 4 weeks and 6 month follow up points. H7: In participants with AD, SAND will be able to assess insight into illness and cognitive function at baseline, and will be able to detect change in insight at follow up points.

ELIGIBILITY:
Inclusion Criteria for AD participants:

1. Age 55 years or above.
2. Ability to understand and speak English.
3. Confirmed Diagnosis of Probable AD by NIA-AA criteria.
4. Either not taking Cognitive enhancers or taking them at a stable dose for the last 3 months.
5. Willingness and ability to provide informed consent or an ability to assent and availability of a substitute decision maker willing to provide consent on participant's behalf.
6. Corrected visual acuity enough to read newspaper headlines.
7. Ability to hear a raised conversational voice, with hearing aids if needed.

Inclusion criteria for healthy control participants:

1. Age 55 or above.
2. Willingness and ability to speak English.
3. Willingness and ability to provide informed consent.
4. Corrected visual acuity enough to read newspaper headlines.
5. Ability to hear a raised conversational voice, with hearing aids if needed.

Exclusion Criteria for AD participants:

1. MOCA score < 10.
2. DSM IV - TR diagnosis of a current episode of mood disorder in the last 3 months.
3. DSM IV - TR diagnosis of a current anxiety disorder in the last 3 months.
4. DSM IV - TR diagnosis of a current substance use disorder in the last 3 months.
5. DSM IV - TR diagnosis of a current or lifetime primary psychotic disorder.
6. Diagnosis of intellectual disability or a neurodevelopmental disorder.
7. Electroconvulsive Therapy treatment in the last 6 months.
8. History of a seizure other than a febrile seizure in infancy.
9. Currently taking Anticonvulsants or Benzodiazepines.
10. Any contraindication for TMS or any other medical condition/circumstances that would make the study participation difficult for the participant.

Exclusion criteria for healthy control participants:

1. Meets criteria for a DSM IV - TR diagnosis other than simple phobias or Adjustment disorder.
2. Any other neurological disorder affecting central nervous system.
3. Psychotropic medication except for sedative /hypnotics at a stable dose for at least 4 weeks.
4. History of seizure other than a febrile seizure in infancy
5. Currently taking Anticonvulsants or Benzodiazepines.
6. Any contraindication for TMS or any other medical condition/circumstances that would make the study participation difficult for the participant.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Change in N-back Task Performance | pre-intervention (baseline) and then 7 days, 4 weeks and 6 months after intervention
  The N-Back is a working memory task where the subject is presented with a sequence of stimuli (letters).
  The task consists of indicating when the current stimulus matches the one from N steps earlier in the sequence. By measuring the accuracy on the N-back task, the investigators will assess the working memory at baseline and compare the change at 7days, 4 weeks and 6 months post-intervention.
  The investigators' pilot data suggests that this test is most discriminatory between AD participants and healthy controls. The N-back task will be administered while recording EEG online to assess theta-gamma coupling.

SECONDARY OUTCOMES:
Changes in Theta Phase-Gamma Amplitude Coupling | Change from baseline at 7 days, 4 weeks and 6 months after intervention.
  Theta gamma coupling may serve as a surrogate marker of neuroplasticity and underlie working memory performance. From EEG recordings, the investigators will assess the changes in this marker from baseline at 7 days, 4 weeks and 6 months after intervention.
Changes in DLPFC Neuroplasticity | Change from baseline at 7 days, 4 weeks and 6 months after intervention.
  The investigators will use a previously established protocol to administer PAS to assess DLPFC neuroplasticity at baseline and compare the changes at 7 days, 4 weeks and 6 months after intervention.
  It involves stimulation on median nerve at wrist followed by TMS of DLPFC after 25 ms delay. PAS-induced neuroplasticity will be measured as the change in TMS-induced cortical evoked activity in response to PAS and as captured with EEG.
Changes in Cognitive Function Measures Scores | Change from baseline at 7 days, 4 weeks and 6 months after intervention.
  The investigators will use an array of neuropsychological (NP) tests to measure the general cognitive functions at baseline and the change from baseline at 7 days, 4 weeks and 6 months after intervention.
  The NP tests include: Executive Interview (EXIT25), Montreal Cognitive Assessment (MOCA) and Cambridge Neuropsychological Test Automated Battery (CANTAB).
Validating a new scale for insight in Alzheimer's disease. | Change from baseline at 7 days and 6 months after intervention.
  The Scale to Assess Anosognosia in Neurocognitive Disorders' (SAND) is a new scale to assess insight in patients with Alzheimer's disease. It measures the core dimensions of clinical insight into AD, including general illness awareness, symptom attribution, awareness of need for treatment, and awareness of negative consequences attributable to the illness.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Kumar, MD, FRCPC, Principal Investigator — Center for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research